CLINICAL TRIAL: NCT03776487
Title: Pilot Study of Dual Checkpoint Inhibition Followed by Immuno-Chemoradiation in Patients With Resectable Gastric Adenocarcinoma (Concept ID 2016-NIV-0551)
Brief Title: Nivolumab, Ipilimumab and Chemoradiation in Treating Patients With Resectable Gastric Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0012; NCI-2018-02344 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0012 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-12-12; First posted 2018-12-14 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Clinical Stage 0 Gastric Cancer AJCC v8; Clinical Stage 0 Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage I Gastric Cancer AJCC v8; Clinical Stage I Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IIB Gastric Cancer AJCC v8; Clinical Stage IIB Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IVA Gastric Cancer AJCC v8; Clinical Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Gastric Adenocarcinoma; Localized Gastric Carcinoma; Localized Gastroesophageal Junction Adenocarcinoma; Pathologic Stage 0 Gastric Cancer AJCC v8; Pathologic Stage 0 Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage I Gastric Cancer AJCC v8; Pathologic Stage IA Gastric Cancer AJCC v8; Pathologic Stage IA Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IB Gastric Cancer AJCC v8; Pathologic Stage IB Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IC Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage II Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIA Gastric Cancer AJCC v8; Pathologic Stage IIA Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIB Gastric Cancer AJCC v8; Pathologic Stage IIB Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIIA Gastric Cancer AJCC v8; Pathologic Stage IIIB Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8
MeSH Terms: interventions — Fluorouracil; dehydroftorafur; Radiotherapy, Intensity-Modulated; Ipilimumab; CTLA-4 Antigen; Nivolumab; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (chemotherapy, immunotherapy, IMRT) (Experimental): INDUCTION CHEMOTHERAPY: Patients receive oxaliplatin IV over 2 hours and fluorouracil IV over 48 hours on day 1. Treatment repeats every 14 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 30 minutes on day 1. Treatment with nivolumab repeats every 2 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Beginning course 4, patients also receive fluorouracil IV continuously for 5 days per week and undergo 25 fractions of IMRT for 5 weeks. Patients undergo surgical resection 5-7 weeks after completing radiation therapy.
  Within 8-12 weeks post-surgery, patients with residual disease may receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 2 weeks for 8 courses (16 weeks) then every 4 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fluorouracil; Radiation: Intensity-Modulated Radiation Therapy; Biological: Ipilimumab; Biological: Nivolumab; Drug: Oxaliplatin; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Procedure: Therapeutic Conventional Surgery — Undergo partial or total gastrectomy and lymphadenectomy

SUMMARY:
This pilot phase I/II trial studies the side effects and how well nivolumab and ipilimumab in combination with chemotherapy and radiation therapy work in treating patients with gastric cancer that can be removed by surgery. Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as oxaliplatin and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Intensity-modulated radiation therapy uses thin beams of radiation of different strengths aimed at the tumor from many angles. This type of radiation therapy may reduce the damage to healthy tissue near the tumor. Giving nivolumab, ipilimumab, chemotherapy and radiation therapy may work better in treating patients with gastric cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and toxicity profile of intravenous nivolumab in combination with ipilimumab after standard chemotherapy and followed by intravenous nivolumab in combination with fluoropyrimidine and intensity-modulated radiation therapy (IMRT) for the treatment of localized gastroesophageal junction (GEJ) and/or gastric cancer.

SECONDARY OBJECTIVES:

I. To assess the efficacy of double checkpoint inhibition (nivolumab + ipilimumab) followed by nivolumab plus chemoradiation.

II. To assess the overall safety and tolerability of adjuvant nivolumab in subjects with resected GEJ or gastric cancer.

III. To evaluate disease free survival (DFS).

IV. To explore changes in tumor stroma profile before and after immunotherapy and radiation therapy.

V. To bank tumor and blood specimen for future correlative analysis, including, but not limited to, biomarker analysis.

OUTLINE:

INDUCTION CHEMOTHERAPY: Patients receive oxaliplatin intravenously (IV) over 2 hours and fluorouracil IV over 48 hours on day 1. Treatment repeats every 14 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 30 minutes on day 1. Treatment with nivolumab repeats every 2 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Beginning course 4, patients also receive fluorouracil IV continuously for 5 days per week and undergo 25 fractions of IMRT for 5 weeks. Patients undergo surgical resection 5-7 weeks after completing radiation therapy.

Within 8-12 weeks post-surgery, patients with residual disease may receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 2 weeks for 8 courses (16 weeks) then every 4 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 and 84 days, every 12 weeks for 2 years, then every 6-12 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have signed and dated an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal subject care. Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.
* All subjects must have localized/eligible for surgery gastric cancer (GC) or GEJ carcinoma type III, with negative peritoneal washing. Subjects must have histologically confirmed predominant adenocarcinoma. The documentation of GEJ involvement can include biopsy, endoscopy, or imaging.
* Subject must be previously untreated with systemic treatment (including HER 2 inhibitors) given as primary therapy for advanced or metastatic disease. No prior neoadjuvant chemotherapy, immunotherapy, radiotherapy and/or chemoradiotherapy are permitted.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Absolute neutrophil count (ANC) >= 1,500/mcL (within 28 days of treatment initiation).
* Platelets >=100,000/mcL (within 28 days of treatment initiation).
* Hemoglobin >= 9 g/dL or > 5.6 mmol/L; if patient is not actively bleeding and has hemoglobin of < 9g/dL, patient can receive blood transfusion to increase hemoglobin to >= 9g/dL (within 28 days of treatment initiation).
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCL]) > 60 mL/min for subjects with creatinine levels > 1.5 x institutional ULN (measured via 24-hour urine collection) (within 28 days of treatment initiation). Creatinine clearance should be calculated per institutional standard.
* Serum total bilirubin =< 1.5 X ULN (1.5 mg/dL or 25.65 umol/L) OR direct bilirubin < ULN for subjects with total bilirubin levels < 1.5 X ULN. Except patients with Gilbert's disease (< 3 X ULN) (within 28 days of treatment initiation).
* Aspartate aminotransferase AST (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR < 5 X ULN for subjects with liver metastases (within 28 days of treatment initiation).
* Albumin >= 3 mg/dL (within 28 days of treatment initiation).
* Prothrombin Time (PT) < 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time PTT is within therapeutic range of intended use of anticoagulants. Activated partial thromboplastin Time (aPTT) < 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (within 28 days of treatment initiation).
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of study drug. Women must not be breastfeeding.
* Prior to chemotherapy and immunotherapy, WOCBP must agree to follow instructions for method(s) of contraception for the duration of study treatment with nivolumab and 5 months after the last dose of study treatment (i.e. 30 days (duration of ovulatory cycle plus the time required for the investigational drug to undergo approximately five half-lives).
* Males who are sexually active with WOCBP must agree to follow instructions for methods of contraception for the duration of study treatment with nivolumab and 7 months after the last dose of study treatment (i.e. 90 days (duration of sperm turnover) plus the time required for the investigational drug to undergo approximately five half-lives). In addition, male subjects must be willing to refrain from sperm donation during this time.

Exclusion Criteria:

* Participants with an active, known or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).

  * NOTE: Testing for HIV must be performed at sites where mandated locally.
* White blood cell (WBC) < 2000/uL.
* Any positive test result for hepatitis B virus or hepatitis C virus indicating presence of virus, e.g. hepatitis B surface antigen (HBsAg Australia antigen) positive, or hepatitis C antibody (anti-HCV) positive (except if hepatitis C virus- ribonucleic acid [HCV-RNA] negative).
* History of allergy or hypersensitivity to study drug components.
* Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
* Patients with serious or uncontrolled medical disorders.
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days
  The Bayesian method of Thall, Simon and Estey will be implemented for toxicity monitoring. Safety data will be summarized using frequency tables by organ system, grade and attribution for the neoadjuvant period and adjuvant period separately.

SECONDARY OUTCOMES:
Response rates | Up to 5 years
  Response rates will be estimated along with the corresponding exact 95% confidence interval.
Incidence of adverse events in patients with resected gastroesophageal junction (GEJ) or gastric cancer | Up to 5 years
  The Bayesian method of Thall, Simon and Estey will be implemented for toxicity monitoring. Safety data will be summarized using frequency tables by organ system, grade and attribution for the neoadjuvant period and adjuvant period separately.
Disease-free survival | From the date of surgery until disease relapse or death, whichever occurred first, assessed up to 5 years
  Will be estimated using the method of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Mariela Blum, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org